CLINICAL TRIAL: NCT06973317
Title: Self-Powered Photodetectors for Smarter Healthcare
Acronym: SPARC
Status: Not yet recruiting | Type: Observational
Sponsor: Wrocław University of Science and Technology (Other)
Collaborators: T. Marciniak Lower Silesian Specialist Hospital in Wrocław (Unknown)
Responsible Party: Principal Investigator, Katarzyna Gwozdz, Principal Investigator, Wrocław University of Science and Technology
Other Study IDs: SPARC
Record Dates: First submitted 2025-05-05; First posted 2025-05-15 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-05

CONDITIONS: Blood Glucose Monitoring
Keywords: Non-invasive monitoring; Photoplethysmography (PPG); Machine learning; Medical devices; glucose

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to evaluate the performance of a novel, non-invasive sensor device based on zirconium oxide photodetector designed to monitor key physiological parameters: blood glucose levels, heart rate, and blood oxygen saturation. The study focuses on adult hospital patients aged 18 to 75, of all sexes, who are undergoing routine monitoring and treatment unrelated to the investigational device.

The main questions this study aims to answer are:

To what extent do the signals obtained from the newly developed device correlate with standard hospital-based methods for measuring blood glucose, heart rate, and blood oxygen saturation?

Is the device feasible, safe, and accurate for use in a real-world clinical setting?

How stable and reproducible are the sensor signals across a demographically diverse patient population?

Can advanced data analysis methods, such as machine learning techniques, be used effectively to interpret the device's output and provide accurate estimates of glucose concentration?

What is the user perception of comfort, safety, and practicality when the device is used in a routine hospital environment?

This study will not assign any interventions to participants; it is purely observational. The novel device is non-invasive, and its use will not interfere with standard clinical care. Measurements will be taken passively or concurrently with routine care procedures.

Participants will:

Continue to receive standard clinical care, including conventional monitoring of glucose, heart rate, and oxygen saturation.

Undergo additional measurements using the investigational device, which will be placed non-invasively on the skin (finger).

Answer a short usability questionnaire assessing their experience with the device, including any discomfort, perceived safety, or ease of use.

Data obtained from the device will be compared with routine clinical data from standard hospital devices (e.g., glucometers, pulse oximeters) to evaluate accuracy and reliability. No pharmacological, radiological, or invasive procedures will be involved.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-75 years
* Able to provide informed consent

Exclusion Criteria:

* Skin diseases or injuries on the fingers (e.g., psoriasis, open wounds, burns)
* Tattoos on the fingers
* Severe peripheral circulation disorders
* Pregnancy
* Presence of active implantable medical devices (e.g., pacemakers)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The populaiton studied will be patients at the Department of Endocrinology, Diabetology and Internal Medicine at the T. Marciniak Lower Silesian Specialist Hospital in Wrocław
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2027-06 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of a Non-Invasive Device for Measuring Blood Glucose, Heart Rate, and Oxygen Saturation | 8 months
  To evaluate the correlation between the signals obtained from the newly developed non-invasive device and standard hospital-based methods for measuring blood glucose levels, heart rate, and blood oxygen saturation. The primary aim is to assess the feasibility, signal stability, and potential accuracy of the investigational device in a clinical setting.

SECONDARY OUTCOMES:
User-friendliness and Practical Usability of the Device in Routine Hospital Procedures | 8 months
  Usability of the device will be assessed using a standardized questionnaire (e.g., System Usability Scale, SUS) completed by clinical staff after performing routine procedures with the device. Additional measures will include the average time (in minutes) required to complete the procedure and the number of use-related errors observed per procedure, recorded by a trained observer.
Variability of Device Readings Across a Demographically Diverse Adult Population | 8 months
  The device's output readings-heart rate (beats per minute), oxygen saturation (%SpO₂), and glucose levels (mg/dL)-will be collected from adult participants aged 18-75, balanced by sex. For each physiological parameter, variability will be assessed using standard deviation and coefficient of variation across repeated measurements. Device readings will be compared to reference standard measurements performed during the patients' routine hospital stay (e.g., laboratory tests) to evaluate consistency.
Applying Machine Learning to Interpret Non-Invasive PPG Signals for Glucose Estimation | 12 months
  To apply and evaluate machine learning techniques for the interpretation of non-invasive PPG signals, in order to estimate glucose levels and benchmark the performance of the sensor platform

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Endocrinology, Diabetology and Internal Medicine at the T. Marciniak Lower Silesian Specialist Hospital in Wrocław, Wroclaw, Lower Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided
Individual Participant Data (IPD) might not be shared for several reasons.
  Firstly, privacy and confidentiality concerns are significant, as even anonymized data could potentially lead to participant identification, especially in smaller datasets. Additionally, legal and regulatory restrictions, such as data protection laws like GDPR, may prevent sharing. Informed consent forms signed by participants might also include clauses that limit data sharing.
  Moreover, data quality and integrity issues could arise if the data is incomplete, inaccurate, or not yet validated for public use. There could also be commercial interests at play, where organizations may consider the data proprietary and choose to restrict access to maintain a competitive advantage. Finally, ethical considerations may arise, as sharing IPD might lead to misuse or misinterpretation of the data outside the intended research scope.